CLINICAL TRIAL: NCT01762488
Title: Renal Denervation in Treatment Resistant Hypertension, a Double-blind Randomized Controlled Trial
Brief Title: Renal Denervation in Treatment Resistant Hypertension
Acronym: ReSET-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Henrik Vase (Other)
Collaborators: Aarhus University Hospital (Other); Regionshospitalet Silkeborg (Other); Randers Regional Hospital (Other); Central Jutland Regional Hospital (Other); Regional Hospital Holstebro (Other)
Responsible Party: Sponsor-Investigator, Henrik Vase, MD, PhD, Aarhus University Hospital Skejby
Organization: Aarhus University Hospital Skejby (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 35218
Record Dates: First submitted 2013-01-04; First posted 2013-01-07 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Hypertension
Keywords: Treatment Resistant Hypertension; Renal Denervation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Renal denervation by ablation of the renal arteries (Active Comparator): By femoral access, renal angiography is performed. The patient will be sedated. In case of acceptable renal artery anatomy allowing renal ablation, the patient will be randomized in the cath. lab. If randomized to active treatment, renal artery ablation will be carried out straight away.
  Interventions: Procedure: Ablation of the renal arteries
- Control (Sham Comparator): By femoral access, renal angiography is performed. The patient will be sedated. In case of acceptable renal artery anatomy allowing renal ablation, the patient will be randomized in the cath. lab. If randomized to sham treatment, the procedure stops.
  Interventions: Procedure: Renal angiography

INTERVENTIONS:
Procedure: Ablation of the renal arteries — Catheter-based renal denervation by applying low power radiofrequency to the renal artery using the EnligHTN Catheter, introduced by femoral artery access.
  Arms: Renal denervation by ablation of the renal arteries
Procedure: Renal angiography — Renal angiography by femoral access
  Arms: Control

SUMMARY:
The purpose of this double-blind, randomized and sham controlled study is to investigate the blood pressure lowering effect of renal denervation by catheter based ablation in the renal arteries in patients with milder forms of treatment resistant hypertension. The effect on blood pressure will be evaluated by 24-hour ambulatory blood pressure measurements at baseline and after 3 and 6 months of follow up. Secondary endpoint evaluation comprises hemodynamic assessment by applanation tonometry and the cold pressor response.

ELIGIBILITY:
Inclusion Criteria:

* Systolic daytime (24 hour-ambulatory blood pressure measurement) > 135 mmHg and < 145 mmHg.
* Stable (for at least 1 month and with no planned changes for the next 6 months) antihypertensive therapy with at least 3 antihypertensive drugs, including a diuretic.
* Documented adherence to present antihypertensive therapy

Exclusion Criteria:

* Pregnancy
* Non compliance
* Heart failure (NYHA Class III-IV)
* LV ejection fraction < 50 %
* Renal insufficiency (eGFR<30 ml/min)
* Unstable coronary heart disease
* Coronary intervention within 6 months
* Myocardial infarction within 6 months
* Claudication
* Orthostatic syncope within 6 months
* Secondary hypertension (except CKD)
* Significant valvular heart disease
* Clinically significant biochemical abnormalities (electrolytes, haemoglobin, hepatic function, thyroid)
* Second and third degree AV block
* Macroscopic haematuria
* Renal artery anatomy not suitable for renal artery ablation (Stenosis, diameter < 4 mm, length < 2 cm or severe calcifications)
* Moderate/severe obstructive sleep apnoea (AHI > 15) if CPAP treatment has not been attempted

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-01; Primary Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in daytime systolic blood pressure (24-hour ambulatory blood pressure measurement) | 6 months

SECONDARY OUTCOMES:
Change from baseline in blood pressure (clinic and 24-hour ambulatory blood pressure measurement) | 3 and 6 months
Change from baseline in central blood pressure, augmentation index and pulse wave velocity | 6 months
Change from baseline in cold pressor response | 6 months
Change from baseline in intensity of medical antihypertensive therapy | 1, 3 and 6 months
Blood pressure (clinic measurement) | 1, 3 and 6 months
Renal function (eGFR and electrolytes) | 1, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Vase, MD, PhD, Study Chair — Skejby Hospital, Dept. of Cardiology
Locations (1):
- Aarhus University Hospital, Skejby, Aarhus, Denmark